CLINICAL TRIAL: NCT02520947
Title: The Effect of BIS Monitorization to Intraoperative Anesthetic and Analgesic Consumption During Coronary Artery Grafting Surgery and Postoperative Mortality and Morbidity
Brief Title: The Effect of BIS Monitorization to Intraoperative Anesthetic Consumption During Coronary Artery Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Ebru Kaval, resident, Baskent University Ankara Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BIS-12345
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Unconscious State
Keywords: desflurane; BIS; coronary artery bypass grafting surgery
MeSH Terms: conditions — Unconsciousness | interventions — Desflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bispectral index (Experimental): The group that desflurane titrated according to bispectral index monitoring
  Interventions: Device: BIS; Drug: Desflurane
- Minimum alveolar concentration (Other): The group that desflurane consumption titrated according to minimum alveolar concentration monitoring
  Interventions: Drug: Desflurane

INTERVENTIONS:
Device: BIS — Bispectral index monitoring
  Other Names: processed electroencephalograpy
  Arms: Bispectral index
Drug: Desflurane — volatile agent for maintenance of anesthesia
  Other Names: suprane

SUMMARY:
213 patients undergoing elective on-pump coronary artery bypass grafting (CABG) were enrolled into this prospective-clinical trial.After hundred and sixty three patients were excluded due to various reasons, 50 patients were randomized to BIS (bispectral index) and MAC (minimum alveolar concentration) groups. In BIS group (Group B, n=25), desflurane was titrated within 40 to 60 BIS values and in MAC group (Group M, n=25) within 0.7 to 1.3 MAC. Primary end point of the study was to investigate the difference of desflurane consumption between groups.

DETAILED DESCRIPTION:
This study was approved by Baskent University Institutional Review Board and Ethics Committee (Project No: KA13/294) and supported by Baskent University Research Fund. The study was conducted in a single university hospital (Başkent University Hospital, Ankara, Turkey). Between January 2014 and October 2014, 213 patients undergoing CABG surgery were assessed for eligibility. 163 patients were excluded because of not meeting inclusion criteria. 50 patients were enrolled into this prospective-clinical trial. All patients were informed of the nature of the study and gave their written consent during preoperative visit performed by the investigators.Diazepam 0.1 mg/kg (Diazem®) and famotidine HCI 40 mg (Famodin®) were given by the oral route to all patients, the day before surgery at 11 pm and midazolam 0.1 mg/kg (Dormicum®) was given to all patients by oral route 30 min before starting anesthesia. After routine 5 lead electrocardiography, pulse oximeter monitoring and peripheric venous and arterial cannulations, endotracheal intubation was performed. BIS monitoring (BIS Quatro Sensor, Aspect Medical Systems, Inc, Norwood, MA, USA) was applied to BIS group in accordance with the manufacturer's instructions. Anesthesia was induced with propofol 1-2 mg/kg and fentanyl 5-7 mcg/kg by intravenous route, based on the patient's physical status. Muscle relaxation was achieved using iv rocuronium 0.6 mg/kg. Desflurane was administered through a calibrated vaporizer (D-Vapor, Drager Medical AG&Co. KG, Lübeck, Germany) in both groups.

In BIS group (Grup B, n=25) desflurane was titrated to maintain a BIS value of 40 to 60. Anesthesia was maintained with remifentanil 0.1-0.4 mcg/kg/min, and desflurane as a volatile agent. In MAC group (Grup M, n=25) desflurane was titrated within 0.7 to 1.3 MAC. During maintenance, all patients were assessed for hypotension (systolic artery pressure (SAP) < 20% from baseline), bradycardia (heart rate (HR) < 45 bpm) or signs of inadequate anesthesia. Inadequate anesthesia was defined as hypertension (SAP >20% from baseline), tachycardia (HR > 100 bpm) or patient movement, eye opening, swallowing, grimacing, lacrimation or sweating. In MAC group, if anesthesia was inadequate, the desflurane concentration was increased in steps of 0.5 vol % as necessary. In BIS group desflurane was titrated for BIS values between 40 and 60. If this was judged insufficient, the infusion rate of remifentanil was increased by 0.05 g/kg/min. Hemodynamic parameters were maintained within 20% of the basal values with dopamine and nitroglycerin, as required. Dopamine was administered 2-20 mcg/kg/min by central venous route. Calcium and noradrenaline were used as iv boluses if needed. All patients were given fluid infusions to maintain central venous pressure between 10-15 mmHg. Hypotension was initially treated with 100-250 mL iv fluid boluses; desflurane concentration was then reduced in steps of 0.5 vol % and finally, an iv vasopressor (dopamine, adrenaline, dobutamine) was given at a dose chosen by the practitioners. Bradycardia was treated with 0.5 mg atropine. Practitioners were reminded of this protocol via a visual protocol in the room. Morphine 0.1 mg/kg was given all of the patients for pain control. The amount of desflurane administered from the start of the anesthesia to the end of surgical procedure was calculated in two groups. The amount of desflurane administered during the procedure was calculated by using the formula below:

Consumption of anesthetic agent in ml/hr = 3 X set concentration % X fresh gas flow L/min.Patient characteristics and surgical variables such as intraoperative blood loss, anesthesia and surgery durations, BIS (bispectral index) and MAC (minimum alveolar concentration) values, intraoperative hemodynamic parameters and drug requirements of patients, amounts of fluid and blood administered, CVP, urine output, features of the surgery were documented by research staff. All patients were transferred to the ICU. Applying an a priory power analysis, 24 patients at least had to be enrolled in each group to detect a reduction of 20% at least in desflurane consumption with a risk of a of 0.05 and a statistical power of 0.8. Vanderbilt University power and sample size calculation program had been used for power analysis.

Data are presented as medians (interquantile ranges), percentages, or number of cases. Continuous data were compared by Mann-Whitney tests. Categorical data were compared with ki-square test. Significance was defined by P values less than 0.05 using a two-tailed test. Data analysis was performed using IBM-SPSS version 20.0 (IBM-SPSS Science Inc., Chicago, IL). Demographic features, intraoperative use of propofol, intraoperative hourly and total amounts of remifentanil, fentanyl, muscle relaxant and morphine, hourly desflurane consumption, hemodynamic parameters, duration of surgery, aortic cross-clamp and cardiopulmonary bypass (CPB) times, defibrillation and pacemaker requirements, maximum positive inotropic and vasodilator drug requirements, amount of intraoperative fluids, blood and blood products used, urine outputs at the end of the surgery and central venous pressure (CVP) values, intraoperative arterial blood gas results were recorded.Durations of intubation, mechanical ventilation, lengths of ICU and hospital stay, 28 days mortality and postoperative complications were also recorded.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing elective on-pump CABG surgery
* Having an American Society of Anesthesiologists' (ASA) physical status of 3 to 4

Exclusion Criteria:

* A contraindication to the administration of the study drugs
* History of psychiatric and/or neurological disorder
* A left ventricular ejection fraction (EF) < 30%
* A body mass index (BMI) > 30 kg/ m2
* Urgent surgery
* Myocard infarction within 48 hours
* Preoperative need for inotropic/vasodilator agents
* History of heart surgery
* Preoperative or intraoperative need for intraaortic balloon pump
* Left ventricular aneurysms
* Severe pulmonary, renal or hepatic dysfunction
* Presence of excessive alcohol intake or drug abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Total and hourly amounts of desflurane consumption | up to 12 hours
  A more than 20 % reduction in total and hourly amounts of desflurane consumption

SECONDARY OUTCOMES:
Time to extubation | up to 2 days
  participants was followed for the duration of extubation
Mortality | 28 days
  participants was followed for 28 days after surgery
Morbidity | 28 days
  participants was followed for 28 days after surgery for any systemic complications